CLINICAL TRIAL: NCT06618638
Title: Clinical Trial for Shared Decision Making Model for Choosing Pharmacotherapy in ADPKD Patients
Brief Title: Shared Decision Making for Choosing Autosomal DOminant Polycystic Kidney Disease Treatment
Acronym: SDM-ADOPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other); Hallym University Kangnam Sacred Heart Hospital (Other); Kangbuk Samsung Hospital (Other); Korea University Guro Hospital (Other); Seoul National University Boramae Hospital (Other); Asan Medical Center (Other); InjeUniversityBusanPaikHospital (Unknown); Chonnam National University Hospital (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HV23C182600
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: ADPKD (autosomal Dominant Polycystic Kidney Disease)
Keywords: Autosomal Dominant Polycystic Kidney Disease; Shared Decision Making; Hybrid Randomized Controlled Trial type 1; Tolvaptan
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SDM group (Experimental): SDM group receives treatment using a shared decision-making model.
  Interventions: Behavioral: Shared decision making model
- Conventional group (Other): Conventional group receives treatment as usual.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Shared decision making model — Shared decision making model for choosing pharmacotherapy in ADPKD patients. This newly developed shared decision making model follows the SHARE approach and includes patient education, identifying values and preferences, reaching a decision and evaluating.
  Arms: SDM group
Behavioral: Usual Care — Usual care for ADPKD patients
  Arms: Conventional group

SUMMARY:
The purpose of this study is to generate clinical evidence and assess the feasibility of a shared decision-making (SDM) model for the selection of Tolvaptan in patients with ADPKD.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) patients, eligible to taking tolvaptan, have to decide whether to take tolvaptan regarding critical factors such as water intake, side effects, and their personal values and preferences. Our study aims to develop and validate a shared decision-making (SDM) model for ADPKD patients considering tolvaptan therapy.

The SDM model we developed include a patient decision aid, educational materials and self-monitoring tools, all provided by a mobile application. This model was built to deliver enough knowledge and considerations during a decision-making process, which would be helpful for patients to reach a decision on tolvaptan.

Through the multi-center hybrid randomized controlled trial, the model's effectiveness and feasibility will be evaluated. Improvements in treatment outcomes, patient satisfaction, adherence, and quality of life are anticipated. This study can propose a structured, patient-centered framework for therapeutic decision-making in ADPKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the age of 18 to 80
* Participants with a diagnosis with CKD stage 2 or 3
* Participants with a diagnosis with ADPKD classified as 1C, 1D, or 1E according to Mayo classification
* Participants with the ability to communicate and use digital devices
* Participants with no severe visual impairment and cognitive dysfunction

Exclusion Criteria:

* Participants who were previously exposured to tolvaptan
* Participants who are contraindicated to tolvaptan
* Participants who were judged ineligible by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in htTKV from baseline to 12 months | From enrollment to the end of treatment at 1 months
  Calculate percent change in height adjusted total kidney volume (htTKV) from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chul Kim, Principal Investigator — Seoul National University Hospital
Locations (9):
- South Korea (9):
  - Hallym University Kangnam Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Republic of Korea
  - InjeUniversityBusanPaikHospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Boramae Hospital, Seoul
  - Korea University Guro Hospital, Seoul